CLINICAL TRIAL: NCT06242210
Title: Effects of Pursed Lip Breathing Technique Versus Stacked Breathing Technique on Dyspnea, Lung Volumes, Oxygenation, and Quality of Life Among Chronic Bronchitis Patients
Brief Title: Effects of Pursed Lip Breathing Technique Versus Stacked Breathing Technique Among Chronic Bronchitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0336
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Bronchitis
Keywords: Pursed Lip Breathing; Stacked Breathing; Dyspnea; Lung Volumes
MeSH Terms: conditions — Bronchitis, Chronic; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pursed Lip Breathing Technique (Experimental): Patient will be asked to attain fowler's position by placing a pillow in front of his trunk to support a comfortable breathing pattern. Then, patient will be instructed to inhale through nose deeply until no more air can be inhaled and which will be followed by a slow expiration through pursed or rounded lip, like at the time of whistling.Patient will also be demonstrated visually for the proper breathing pattern even for once to multiple times till complete understanding before performing itself. The technique will be administered to the patient under supervision for 10 minutes, and the patient will be instructed to use this trained exercise in his daily routine as per needed.
  Interventions: Other: pursed lip
- Stacked Breathing (Experimental): Patient will be asked to attain recumbent position by lying supine at a reclining angle to support a comfortable breathing pattern. Then, patient will be instructed to inhale slowly and deeply once through nose and hold it, then inhale again slowly and deeply through nose and trap the air in again over the first one, then inhale again until no more air can be inhaled and which will be held for a bit then followed by a slow and quiet expiration. Patient will also be demonstrated visually for the proper breathing pattern even for once to multiple times till complete understanding before performing itself
  Interventions: Other: Stacked Breathing

INTERVENTIONS:
Other: pursed lip — pursed lip breathing technique for group A through videos on smart phones and a brochure given to patients. Each session takes 15-20 minutes until researchers ensure that patients understand how to perform exercises and re-demonstrate them. • Each group applied it twice per day for a period of 4 weeks. Telephone follow-up was used for patients in both groups
  Arms: Pursed Lip Breathing Technique
Other: Stacked Breathing — The technique will be administered to the patient under supervision for 10 minutes, and the patient will be instructed to use this trained exercise in his daily routine as per needed
  Arms: Stacked Breathing

SUMMARY:
Chronic bronchitis is a non-allergic, inflammatory disease that is developed because of inflamed bronchial walls, and, is characterized by persistent cough with sputum for 3 months for 2 consecutive years at least. It affects males more than females at the age of 40 years, with increasing incidence as the age progresses. Chronic bronchitis is associated with multiple health-related issues like; dyspnea, reduced lung volumes and capacities, poor quality of life, and physical inactivity. Its clinical manifestations are coped with using the pharmaceutical approach, surgical maneuvers, and pulmonary rehabilitation. In the context of pulmonary rehabilitation, pursed lip breathing and stacked breathing are evident to deal with symptoms of chronic bronchitis and make the individuals lead a physically active and healthy life. In this research study, patients will be enrolled with strict adherence to eligibility criteria and then allocated into two groups by using the convenience sampling technique after having their written informed consent form. The participants will either receive pursed lip breathing technique or a stacked breathing technique, which will be followed by baseline treatment at every session. Both groups will be then subjected to receive intervention that will take a duration of 40 minutes every session, 30 minutes of baseline treatment, and 10 minutes of intervention, for the period of 2 weeks with the frequency of performing the intervention thrice per day. The outcomes will be evaluated by using a modified Borg scale for dyspnea, a peak expiratory flow meter for lung volumes, a pulse oximeter for oxygenation, and EuroQol; 5D-5L for quality of life. Data will be recorded at pre-treatment, on the 1st day, and post-treatment, on the 14th day. The recorded data will be then entered and analyzed using SPSS (Statistical Package of Social Sciences) version 23.

ELIGIBILITY:
Inclusion Criteria:

* Both genders will be included.
* Patients lie in the age ranges from 40 to 60 years.
* Patients diagnosed with chronic bronchitis. for more than one year.
* Patients presents with reduction in movements of chest wall, which reduces the area of entrance for air.
* Patients who have no history of usage of corticosteroids and anabolic steroid from previous three months.
* Patients do not experience severe obstruction of airflow i.e.: value of FEV1 is at 50% of the predicted value.
* Patients have no history or persistence of COVID-19

Exclusion Criteria:

* • Any recent thoracic surgeries and abdominal surgeries.

  * Patients lie at the Grade IV of modified medical research council dyspnea scale.
  * Patients who present with history of any respiratory disease from two preceding months.
  * Patients receiving any maneuvers of pulmonary rehabilitation from previous two months.
  * Patients who experience chronic respiratory failure demanding for supplemental oxygen.
  * Patients have persisting cardiac and pulmonary hypertension that interferes with compliance of intervention.
  * Patients who had other chronic respiratory diseases, new or current smoker, and had respiratory tract infection

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Modified Borg Scale | baseline and fourth week
  The Modified Borg Dyspnea Scale has demonstrated both validity and reliability in various populations, including both healthy individuals and clinical patients with a highly significant values of Pearson's correlation coefficient and Spearman's correlation coefficient that lies within the range of 0.5 to 0.99, which showsa p-value of less than 0.05. Its ease of use has made it widely employed for monitoring exercise intensity in exercise prescription and rehabilitation settings
Spirometer | baseline and fourth week
  Spirometry is a maneuver that works on the principle of forced expiration, and is constituted of FEV1; that signifies the volume of air pushed out of lung forcefully within one second, FVC; which represents the forced vital capacity of lungs and ratio of FEV1 / FVC, to measure the limitation faced by patients of chronic bronchitis during airflow. Spirometry is considered to be a gold standard instrument that has been employed to assess the forced expiratory flow parameters among patients of COPD, asthma, chronic bronchitis. It been proven to be a highly reliable and valid tool on the basis of value of 95% confidence interval that was determined from 0.51 to 0.86, with the purpose to keep lung volumes under surveillance
Pulse Oximeter | baseline and fourth week
  Healthcare professionals worldwide use pulse oximeter on a daily basis to obtain a noninvasive measurement of SpO2, which reflects arterial oxygen saturation (SaO2). This measurement aids in identifying and addressing hypoxemia (low oxygen levels) and hyperoxemia (high oxygen levels). Pulse oximetry monitoring is commonly regarded as the fifth vital sign and is particularly recommended for patients in need of oxygen therapy
European Quality of Life; 5 Dimensions, 5 Levels Questionnaire | baseline and fourth week
  The EQ-5D-5L includes a descriptive system consisting of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with one item per dimension. By assigning preference-based weights (usually specific to each country), the responses to these items can be converted into a single measure of health utility. Furthermore, the instrument provides instructions for indicating overall health status of present day on a visual analog scale.EuroQol;5D-5L is a valid and reliable tools with inter-rater correlation coefficient value of 0.7, and a value of convergent validity of 0.756 under the domain of Spearman Rho Rank correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Younis, MSPT (CP), Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkatesan P. GOLD COPD report: 2023 update. Lancet Respir Med. 2023 Jan;11(1):18. doi: 10.1016/S2213-2600(22)00494-5. Epub 2022 Nov 30. No abstract available. PMID 36462509
- [Background] Mayr AK, Valipour A. Modern Bronchoscopic Treatment Options for Patients with Chronic Bronchitis. J Clin Med. 2023 Feb 26;12(5):1854. doi: 10.3390/jcm12051854. PMID 36902641
- [Background] Satia I, Mayhew AJ, Sohel N, Kurmi O, Killian KJ, O'Connell ME, O'Byrne PM, Raina P. Language and geographical location influence the incidence of chronic cough in the Canadian Longitudinal Study on Aging. ERJ Open Res. 2022 Feb 21;8(1):00721-2021. doi: 10.1183/23120541.00721-2021. eCollection 2022 Jan. PMID 35198625